CLINICAL TRIAL: NCT00665132
Title: Acute Human Study: StimRouter for Peripheral Nerve Stimulation of Discrete Peripheral Nerves
Acronym: StimRouter
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bioness Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-STMR07-001-Rev A.1
Record Dates: First submitted 2008-04-21; First posted 2008-04-23 (Estimated); Results first posted 2016-06-06 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-05

CONDITIONS: Unilateral Carpal Tunnel Syndrome
Keywords: wrist; hand; pain; failed CTR; carpal tunnel syndrome; CTS; CTR; carpel tunnel release; Peripheral nerve; Median nerve
MeSH Terms: conditions — Pain; Carpal Tunnel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- StimRouter (SR) for CTS (Experimental): Percutaneous implantation of StimRouter System
  Interventions: Device: StimRouter System

INTERVENTIONS:
Device: StimRouter System — Implanted with StimRouter System receive 6 hours (or less if not tolerated by the Subject)of electrical therapeutic stimulation each day for a total of 5 days (from start of successful programming)

SUMMARY:
This study is being done to see how well a new investigational medical device, the StimRouter (STR) System, will work to treat the chronic pain in people who have failed previous treatments for Carpal Tunnel Syndrome (CTS) pain, including surgery. These people have been treated for CTS pain before including surgical carpal tunnel release, but without good results, and they are still having pain. The study will look at both the good and bad effects of the StimRouter System for treating this kind of pain and as a general peripheral nerve stimulation device for treating chronic pain. The study will also help to understand other possible uses for the StimRouter System.

DETAILED DESCRIPTION:
This is a prospective, single-center, open label study designed to evaluate the clinical use of the StimRouter (STR) as a peripheral nerve stimulation device for the treatment of chronic pain. The clinical study is proposed to serve as an evaluation of the preliminary StimRouter design, proposed implantation techniques, electrical stimulation parameters, and outcome measures for the StimRouter. The current study will utilize the median nerve (in the context of carpal tunnel syndrome (CTS), status-post a single failed carpal tunnel release (CTR) surgery)as a model to represent the device's more general intended use as a peripheral nerve stimulator to treat chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Chronic peripheral pain persisting for greater than or equal to 3 months diagnosed previously as a mononeuropathy of the median nerve at the level of the carpal tunnel (i.e., diagnosed CTS)
* Average chronic pain level greater than or equal to 5/10 [on 0-10 numeric rating scale (NRS) (BPI#14)], where such pain is attributed to injury, irritation, or entrapment of the median nerve at the level of the carpal tunnel (i.e., diagnosed CTS)
* Failure of a single prior carpal tunnel release surgery to provide relief, where such failed surgery was performed greater than or equal to study entry
* Able to tolerate stimulation (TENS)
* Temporary pain relief is achieved by local anesthetic block of the target median nerve suspected to be the source of chronic pain symptoms
* Ability to give informed consent and understand study requirements
* Ability to quantify pain using a 0-10 numeric rating scale [A screening tool will be used to ensure that subjects can rate 3 common pain scenarios (mosquito bite, stubbed toe and broken bone) on a 0-10 NRS relative to each other, with mosquito bite < stubbed toe < broken bone]
* Willing and able to understand and comply with all study-related procedures during the course of the study
* Motivated to maintain an accurate diary for the study duration

Exclusion Criteria:

* Metal implants in the forearm
* Active infection
* Active or existing skin disorder or irritation which, at the physician's discretion, contraindications use of skin gel electrodes
* Allodynia
* Regular use of antiplatelet medications [e.g., aspirin, ticlopidine (Ticlid), clopidogrel (Plavix), tirofiban (Aggrastat), and eptifibatide (Integrilin)]
* Anticoagulated (taking warfarin or heparin, including fractionated heparin) or has a bleeding disorder
* Cardiac pacemaker
* Implanted neurostimulator (e.g., spinal cord, deep brain, vagus nerve stimulator) or implanted pump or infusion device
* History of cardiac arrhythmia with homodynamic instability
* Untreated drug habituation or dependence
* Psychologically or medically unstable
* Uncontrolled seizures (averaging > 2 seizures per month)
* Pregnant or plan on becoming pregnant or breastfeeding during the study period
* Currently require, or likely to require, diathermy and/or MRI during the study duration
* History of adverse reactions to local anesthetic (e.g., lidocaine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-04; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evan L. Rosenfeld, MD, JD, Study Director — Bioness Inc
Locations (1):
- The Center for Pain Relief, Charleston, West Virginia, United States

REFERENCES:
- [Background] Eisenberg E, Waisbrod H, Gerbershagen HU. Long-term peripheral nerve stimulation for painful nerve injuries. Clin J Pain. 2004 May-Jun;20(3):143-6. doi: 10.1097/00002508-200405000-00003. PMID 15100589
- [Background] Day M. Neuromodulation: spinal cord and peripheral nerve stimulation. Curr Rev Pain. 2000;4(5):374-82. doi: 10.1007/s11916-000-0021-7. PMID 10998746

RESULTS

PARTICIPANT FLOW:
Groups:
- StimRouter Stimulation: Percutaneous implantation of StimRouter System
  StimRouter System: Patient is Implanted with StimRouter System lead and receive approximately 6 hours of electrical therapeutic stimulation each day for a total of 5 days (from start of successful programming).
Period: Overall Study
Arm/Group | StimRouter Stimulation
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 1. >/=18 years of age
  2. Carpal Tunnel chronic peripheral pain >/=3 mo with mean pain >/=5/10
  3. Failed prior carpal tunnel release surgery >/=3 mo
  4. Tolerates transcutaneous electrical nerve stimulation (TENS)
  6. Pain relief by local anesthetic block of target nerve 7. Give informed consent 8. Quantify pain using 0 to 10 NRS
Groups:
- StimRouter (SR) Active Stimulation: Percutaneous implantation of StimRouter System
  StimRouter System: Implanted with StimRouter System receive approximately 6 hours of electrical therapeutic stimulation each day for a total of 5 days (from start of successful programming).
Arm/Group | StimRouter (SR) Active Stimulation
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10
Average pain level [Mean (Standard Deviation); unit: units on a scale] — Brief Pain Inventory (BPI) is an 11-point numerical rating scale (NRS) used to rate pain intensity, where zero (0) indicates ''no pain'' and 10 indicates ''pain as bad as you can imagine.'' At enrollment, participants circled the number that best described how much baseline pain they had 'on average' (mean score).
  units on a scale | 6.7 (1.6)

OUTCOME MEASURES:

1. Primary Outcome: Implant Success
Description: Success of device implantation was defined as uncomplicated minimally-invasive implantation of the StimRouter Lead near the targeted peripheral median nerve, resulting in production of desired paresthesias in the sensory distribution of the median nerve when active peripheral nerve stimulation was applied. This outcome parameter was intended to serve as an indication that the lead and electrode stimulating positions could be correctly placed while still maintaining the minimal invasiveness of the procedure. Fluoroscopic imaging was used to document positioning of the StimRouter Lead and, by applying stimulation from a commercially available Dakmed External Pulse Generator (EPG) to the StimRouter Lead, desired paresthesia response was confirmed.
Time Frame: at device implantation procedure
Measure: Number; unit: participants with successful implant
Arm/Group | StimRouter (SR) Active Stimulation
Number analyzed (Participants) | 10
participants with successful implant | 10

2. Secondary Outcome: Patent Satisfaction
Description: Numerical rating scale (NRS) of 0-10 where 0 = not satisfied and 10 = very satisfied
Time Frame: Day 5 after final stimulation
Population: All ten subjects responses were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | StimRouter (SR) Active Stimulation
Number analyzed (Participants) | 10
units on a scale | 9.6 (0.7)

3. Secondary Outcome: Percent of Participants Reporting Pain Change From Baseline to Day 5
Description: Brief Pain Inventory (BPI) questions 14 and 15 were used to measure pain change after 5 days use of StimRouter System. In the BPI, an 11-point numerical rating scale (NRS) is used to rate pain intensity, where zero (0) indicates ''no pain'' and 10 indicates ''pain as bad as you can imagine.'' At enrollment, participants circled the number that best described how much baseline pain they had 'on average' (BPI #14). After enrollment and during the study, patients circled the one number that best described how much pain they had at that time 'right now' (BPI #15). The percent of participants with change from Baseline to Day 5 was calculated.
Time Frame: Day 5
Population: All ten participants were analyzed.
Measure: Number; unit: percentage of patients
Arm/Group | StimRouter (SR) Active Stimulation
Number analyzed (Participants) | 10
percentage of patients | 90

4. Secondary Outcome: Mean Change in Pain Achieved by Participants Who Reported Pain Change From Baseline to Day 5
Description: Using Brief Pain Inventory questions 14 and 15, those 9 subjects who had pain change from Baseline to Day 5 were analyzed to determine change in pain for the overall group. In the BPI, an 11-point NRS is used to rate pain intensity, with a 0 for ''no pain'' and a 10 for ''pain as bad as you can imagine.'' At Baseline, patients circled the number that best described how much baseline pain they had 'on average' (BPI #14). During the study, patients circled the one number that best described how much pain they had at the time 'right now' (BPI #15).
Time Frame: Day 5 after final stimulation
Population: Nine subjects who reported change after 5 days of StimRouter System use are analyzed to determine mean change in pain from Baseline to Day 5 of Stimulation for the overall group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | StimRouter (SR) Active Stimulation
Number analyzed (Participants) | 9
units on a scale | 2.9 (2.0)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from screening throughout the five days of StimRouter stimulation.
Arm/Group | StimRouter (SR) Active Stimulation
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 3/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | StimRouter (SR) Active Stimulation (N=10)
Throbbing in arm (Musculoskeletal and connective tissue disorders) | 1 (1) — Non-device related throbbing in arm after screening visit was mild transient and resulted on no sequelae.
allergic reaction to antiseptic (Immune system disorders) | 1 (1) — Non-device related Bacitracin reaction
Seizure (Nervous system disorders) | 1 (1) — non-device related seizure prior to device implantation procedure

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less